CLINICAL TRIAL: NCT01977261
Title: High Tibial Osteotomy for Osteoarthritis of the Knee: a Randomised Controlled Trial
Brief Title: High Tibial Osteotomy for Osteoarthritis of the Knee
Acronym: HTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, T. Duivenvoorden, M.D., Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2001-HTO
Record Dates: First submitted 2013-10-25; First posted 2013-11-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Opening-wedge HTO (Experimental): Opening-wedge high tibial osteotomy fixated with a Puddu-plate
  Interventions: Procedure: Opening-wedge HTO
- Closing-wedge HTO (Active Comparator): Closing-wedge high tibial osteotomy fixated with 2 staples
  Interventions: Procedure: Closing-wedge HTO

INTERVENTIONS:
Procedure: Opening-wedge HTO — Opening-wedge high tibial osteotomy fixated with a Puddu plate
  Other Names: open wedge high tibial osteotomy
  Arms: Opening-wedge HTO
Procedure: Closing-wedge HTO — Closing-wedge high tibial osteotomy fixated with two staples
  Other Names: Closed wedge high tibial osteotomy
  Arms: Closing-wedge HTO

SUMMARY:
A prospective, randomised, controlled trial compared two different techniques of high tibial osteotomy with a lateral closing wedge or a medial opening wedge, stabilised by a Puddu plate. The clinical outcome and radiological results were examined at one year.

DETAILED DESCRIPTION:
A prospective, randomised, controlled trial compared two different techniques of high tibial osteotomy with a lateral closing wedge or a medial opening wedge, stabilised by a Puddu plate. The clinical outcome and radiological results were examined at one year.

The primary outcome measure was the achievement of an overcorrection of valgus of 4°. Secondary outcome measures were the severity of pain (visual analogue scale), knee function (Hospital for Special Surgery score), and walking distance.

ELIGIBILITY:
Inclusion Criteria:

* Radiological OA, medial joint pain and varus malalignment

Exclusion Criteria:

* Symptomatic OA of the lateral compartment, rheumatoid arthritis, ROM <100, collateral ligament laxity, history of fracture of previous open operation of the lower limb and a flexion contracture > 10 degrees.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2001-01; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
The achievement of an overcorrection of valgus of 4°. | one year
  The achieved correction will be determined on a whole leg radiograph.

SECONDARY OUTCOMES:
Severity of pain | one year
  Severity of pain will be measured with the visual analogue scale
Knee function | one year
  Knee function will be measured with the Hospital for Special Surgery score
Walking distance | one year

OTHER OUTCOMES:
Number of participants with adverse events | one year
  Number of participants with adverse events; infection, loss of correction, hardware removal, implant failure, pseudoarthrosis, peroneal nerve injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Centre, Rotterdam, Netherlands